CLINICAL TRIAL: NCT02481258
Title: A Phase II Randomized, Placebo-Controlled, Double-Blinded Study Evaluating the Effects of Ataciguat (HMR1766) on Aortic Valve Calcification in Patients With Moderate Calcific Aortic Valve Stenosis
Brief Title: A Study Evaluating the Effects of Ataciguat (HMR1766) on Aortic Valve Calcification
Acronym: CAVS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Sanofi (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jordan D. Miller, Ph.D., SAC II, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 14-006469; TR 000954 (Other: National Center for Advancing Translational Sciences)
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Aortic Valve Stenosis
Keywords: Stenosis; Aortic Valve; Aorta; Calcified; Calcific; Calcification
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic; Calcinosis | interventions — 5-chloro-2-(5-chlorothiophene-2-sulfonylamino)-N-(4-(morpholine-4-sulfonyl)phenyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ataciguat (HMR1766) (Experimental): 200mg taken daily for 12 months
  Interventions: Drug: Ataciguat (HMR1766)
- Matching Placebo (Placebo Comparator): Taken Daily for 12 months
  Interventions: Other: Placebo Comparator: Matching Placebo

INTERVENTIONS:
Drug: Ataciguat (HMR1766)
  Arms: Ataciguat (HMR1766)
Other: Placebo Comparator: Matching Placebo
  Arms: Matching Placebo

SUMMARY:
The primary objective of the current study is to determine whether Ataciguat (HMR1766) slows progression of valve calcification in patients with moderate calcific aortic valve stenosis. Secondary and tertiary objectives are to determine whether Ataciguat slows progression of aortic valve function, reduces systemic inflammation, and prevents left ventricular dysfunction in patients with moderate calcific aortic valve stenosis.

DETAILED DESCRIPTION:
Patients with Moderate Calcific Aortic Valve Stenosis may be eligible for enrollment in this study. Participation lasts 12 months, which includes a total of 3 study visits (baseline/screening visit, 6 month follow up visit and 12 month follow up visit). During each visit, a blood sample will be taken along with other research related tests (Orthostatic Tolerance Standing Test, CT Scan, Echocardiogram, DEXA Scan). Qualifying Participants will be supplied with 6 months worth of study medication or placebo during visits 1 (baseline/screening visit) and 2 (6 month follow up visit) in which they will take at home daily with food. On visit 3 (12 month follow up visit), any remaining study medication or placebo will be returned to study staff.

ELIGIBILITY:
Inclusion Criteria

1. Age > 50 years
2. Male or female sex
3. Aortic valve area greater than 1.0 cm2 but less than 2.0 cm2
4. Aortic valve calcium levels greater than 300 AU from chest CT
5. Ejection fraction >50%

Exclusion Criteria

1. Orthostatic intolerance or symptomatic hypotension prior to study or during study visits
2. Positive pregnancy test during screening visit
3. Nitrate use or α-antagonist medication use within 24 hours
4. Systolic blood pressure <110 mm Hg
5. Mean systemic arterial pressure <75 mm Hg
6. Severe mitral or aortic regurgitation
7. Retinal or optic nerve problems
8. Recent (≤30 days) acute coronary syndrome
9. Oxygen saturation <90% on room air
10. Congenital valve disease
11. Hepatic dysfunction/elevated liver enzymes
12. Prescription of drugs known to alter NO-sGC-cGMP signaling (sildenafil, nitrates, etc.)
13. Prescription of Warfarin (Coumadin) for chronic anticoagulation
14. Concomitant participation in other trials at Mayo Clinic or elsewhere
15. Use of phenytoin or related compounds for any indication
16. Chronic midazolam treatment for any indication
17. Use of monoamine oxidase inhibitors for any indication
18. Use of anti-diabetic drugs in the sulfonylurea family

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D Miller, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Zhang B, Enriquez-Sarano M, Schaff HV, Michelena HI, Roos CM, Hagler MA, Zhang H, Casaclang-Verzosa G, Huang R, Bartoo A, Ranadive S, Joyner MJ, Pislaru S, Nkomo VT, Kremers WK, Araoz PA, Singh G, Walters MA, Hawkinson J, Cunningham KY, Sung J, Dunagan B, Ye Z, Miller JD. Reactivation of Oxidized Soluble Guanylate Cyclase as a Novel Treatment Strategy to Slow Progression of Calcific Aortic Valve Stenosis: Preclinical and Randomized Clinical Trials to Assess Safety and Efficacy. Circulation. 2025 Apr;151(13):913-930. doi: 10.1161/CIRCULATIONAHA.123.066523. Epub 2025 Feb 24. PMID 39989354
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were required to complete initial testing for valve calcium and function (in addition to other tests/screening characteristics) prior to enrollment.
Groups:
- Ataciguat (HMR1766): 200mg taken daily for 6 months
  Ataciguat (HMR1766)
- Matching Placebo: Taken Daily for 6 months
  Placebo Comparator: Matching Placebo
Period: Overall Study
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ataciguat (HMR1766): 200mg taken daily for 12 months
  Ataciguat (HMR1766)
- Matching Placebo: Taken Daily for 12 months
  Placebo Comparator: Matching Placebo
- Total: Total of all reporting groups
Arm/Group | Ataciguat (HMR1766) | Matching Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (4) | 72 (8) | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrollment was confined to patients able to travel to Mayo Clinic Rochester for a minimum of 2 visits (baseline/6mo and potentially 12mo)
  Participants
    United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Changes in Aortic Valve Calcium Levels
Description: This will be done using computed tomography (CT) scanning to evaluate aortic valve calcium levels, which is considered to be a "gold standard" for evaluating valvular calcium burden. As measured in Arbitrary Units (AU).
Time Frame: baseline, 6 mos
Measure: Mean (Standard Error); unit: Arbitrary Units
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Number analyzed (Participants) | 12 | 12
Arbitrary Units | 65 (45) | 215 (58)
Statistical Analysis 1: Comparison: Ataciguat (HMR1766) vs Matching Placebo; The statistical analysis was done using an ANCOVA analysis adjusting for the baseline aortic valve calcium levels; Test type: Equivalence — Power calculations were based on a two-sample t-test. A priori calculations to detect an effect size of 0.57 units indicated that that 50 patients per arm were needed to have 80% power. The actual effect size observed in the present study was 0.86; p = 0.05, ANCOVA

2. Secondary Outcome: Change in Levels of Plasma Interleukin-6
Description: Determine whether long-term treatment with HMR1766 will result in sustained increases in systemic sGC signaling and reduce levels of circulating inflammatory cytokines in patients with mild to moderate CAVS. This will be done using ELISA-based measurements of interleukin-6 and tumor necrosis factor alpha in venous blood samples. Key comparisons will be between HMR1766-treated and placebo-treated groups, where we will examine the change in inflammatory cytokine levels from baseline in subjects receiving HMR1766 or placebo capsules.
Time Frame: baseline, 6 mos
Population: One placebo sample was not obtained/available for analysis, thereby reducing the number of data points from 11 to 10.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Number analyzed (Participants) | 12 | 10
pg/ml | 2.3 (1.6) | -0.2 (0.4)

3. Secondary Outcome: Change in Aortic Valve Function: Aortic Valve Area
Description: Determine whether long-term treatment with HMR1766 will result in sustained increases in systemic sGC signaling slow progression of aortic valve dysfunction in patients with mild to moderate CAVS. This will be done using echocardiography-based measurements of aortic valve function. Key comparisons will be between HMR1766-treated and placebo-treated groups, where we will examine the change in:
  1. aortic valve area over time (calculated from the continuity equation) in subjects receiving HMR1766 or placebo capsules, AVA will be evaluated by both the absolute value and following normalization for body surface area, and
  2. mean transvalvular pressure gradient over time (calculated from the blood velocity trace using the Bernoulli equation) in subjects receiving HMR1766 or placebo capsules.
Time Frame: baseline, 6 mos
Measure: Mean (Standard Error); unit: change in cm^2
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Number analyzed (Participants) | 12 | 11
change in cm^2 | -0.07 (0.03) | -0.129 (0.04)
Statistical Analysis 1: Comparison: Ataciguat (HMR1766) vs Matching Placebo; Test type: Equivalence — Power calculations were based on a two-sample t-tests assuming initial recruitment of 50 subjects; p > 0.05, ANCOVA — Our a priori threshold for statistical significance was p < 0.05

4. Secondary Outcome: Change in Left Ventricular Function
Description: Determine whether long-term treatment with HMR1766 will result in sustained increases in systemic sGC signaling slow progression of aortic valve dysfunction in patients with mild to moderate CAVS. This will be done using echocardiography-based measurements of aortic valve function. Key comparisons will be between HMR1766-treated and placebo-treated groups, where we will examine the change in: 1. Left ventricular systolic function (measured by echocardiographic measurement of left ventricular ejection fraction) and 2. Left ventricular diastolic function (measured using the E/A ratio derived from Doppler measurements).
Time Frame: baseline, 6 mos
Measure: Mean (Standard Error); unit: percent
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Number analyzed (Participants) | 12 | 11
percent | 0.6 (1.5) | -2.8 (1.6)
Statistical Analysis 1: Comparison: Ataciguat (HMR1766) vs Matching Placebo; The statistical analysis was done using an ANCOVA analysis adjusting for the baseline aortic valve calcium levels; Test type: Equivalence — Power calculations were based on a two-sample t-test; p > 0.05, ANCOVA — Our a priori threshold for statistical significance was p < 0.05

5. Secondary Outcome: Change in Plasma Tumor Necrosis Factor Alpha
Description: Determine whether long-term treatment with ataciguat reduces levels of circulating inflammatory cytokines.
Time Frame: Baseline, 6 months
Population: One placebo sample was not obtained/available for analysis, thereby reducing the number of data points from 11 to 10.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Number analyzed (Participants) | 12 | 10
pg/ml | 1.9 (2.3) | 2.8 (1.9)

6. Secondary Outcome: Change in Aortic Valve Function: Transvalvular Pressure Gradient
Description: as for outcome 3
Time Frame: baseline, 6 mos
Measure: Mean (Standard Error); unit: change in mm Hg
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
Number analyzed (Participants) | 12 | 11
change in mm Hg | 1.8 (0.85) | 3.6 (0.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were acquired during the periods of patient enrollment (from 6 months to a maximum of 12 months of treatment duration). The total study duration was 3 years.
Description: Our definitions of AE and SAE do not differ from those provided on clinicaltrials.gov. For this study, adverse events were identified through regularly scheduled follow-up phone calls by study staff.
Arm/Group | Ataciguat (HMR1766) | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 1/12
Other Adverse Events (participants affected / at risk) | 9/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ataciguat (HMR1766) (N=12) | Matching Placebo (N=12)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0) — Elevated liver enzymes at 6 month follow-up with clinically-indicated testing showing hepatic inflammation. Resolved after discontinuation of study drug. Not definitive whether hepatotoxicity was due to study drug or other medications taken.
Hospitalization due progression of disease (Cardiac disorders) | 0 (0) | 1 (1) — Patient reported to the hospital with dyspnea and fatigue. Subsequent testing revealed that patient had progressed to severe aortic valve stenosis during the follow-up period and was deemed eligible for surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ataciguat (HMR1766) (N=12) | Matching Placebo (N=12)
Headache (Nervous system disorders) | 0 (0) | 2/11 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Dizziness/Lightheadedness (Nervous system disorders) | 2 (6) | 3 (3)
Nosebleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rash/Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tired/Fatigue (Nervous system disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Odor in urine (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain/Tightness (Cardiac disorders) | 2 (2) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mood Changes (Nervous system disorders) | 1 (1) | 1 (1)
Ankle Edema (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fall (study unrelated) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject tripped and fell. No sustained injuries as a result.
Runny Nose (Common Cold) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot Flashes (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Nervous system disorders) | 1 (1) | 1 (1)
Prostate Cancer (study unrelated) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholesterol lab values out of range (Hepatobiliary disorders) | 0 (0) | 1 (1)
Muscle Cramps/Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (related to cold/flu) (Infections and infestations) | 1 (1) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arm Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT02481258/Prot_SAP_000.pdf